CLINICAL TRIAL: NCT03012854
Title: Different Surgical Procedures of Peroral Endoscopic Myotomy(POEM) for Esophageal Achalasia: a Multicenter Prospective Randomized Controlled Trial
Brief Title: Different Surgical Procedures of Peroral Endoscopic Myotomy(POEM) for Esophageal Achalasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Wei Gong, Doctor of Medicine，Associate Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NFEC-2016-186
Record Dates: First submitted 2017-01-05; First posted 2017-01-06 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Esophageal Achalasia; Esophageal Motility Disorders
Keywords: Esophageal achalasia; Peroral endoscopic myotomy; POEM
MeSH Terms: conditions — Esophageal Achalasia; Esophageal Motility Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- short-myotomy (Experimental): Short-POEM for patients with esophageal achalasia
  Interventions: Procedure: short-myotomy
- long-myotomy (Active Comparator): Long-POEM for patients with esophageal achalasia
  Interventions: Procedure: long-myotomy
- full-thickness myotomy (Experimental): Full-thickness-POEM for patients with esophageal achalasia
  Interventions: Procedure: full-thickness myotomy
- circular myotomy (Active Comparator): Circular-POEM for patients with esophageal achalasia
  Interventions: Procedure: circular myotomy

INTERVENTIONS:
Procedure: short-myotomy — 1. Entry to submucosal space. After submucosal injection, a 2-cm longitudinal mucosal incision is made at approximately 8-10 cm proximal to the gastroesophageal junction (GEJ).
  2. Submucosal tunnelling. A long submucosal tunnel is created to 3 cm distal to the GEJ.
  3. Endoscopic myotomy is carried out in a proximal to distal direction to a total length less than 7 cm. The expected end point of myotomy is 2 cm distal to the GEJ.
  4. Myotomy of inner circular muscle bundles and outer longitudinal muscle layer is done.
  5. Closure of mucosal entry: the mucosal incision is closed using hemostatic clips.
  Arms: short-myotomy
Procedure: long-myotomy — 1. Entry to submucosal space. After submucosal injection, a 2-cm longitudinal mucosal incision is made at approximately 8-10 cm proximal to the gastroesophageal junction (GEJ).
  2. Submucosal tunnelling. A long submucosal tunnel is created to 3 cm distal to the GEJ.
  3. Endoscopic myotomy is carried out in a proximal to distal direction to a total length more than 7 cm. The expected end point of myotomy is 2 cm distal to the GEJ.
  4. Myotomy of inner circular muscle bundles and outer longitudinal muscle layer is done.
  5. Closure of mucosal entry: the mucosal incision is closed using hemostatic clips.
  Arms: long-myotomy
Procedure: full-thickness myotomy — 1. Entry to submucosal space. After submucosal injection, a 2-cm longitudinal mucosal incision is made at approximately 8-10 cm proximal to the gastroesophageal junction (GEJ).
  2. Submucosal tunnelling. A long submucosal tunnel is created to 3 cm distal to the GEJ.
  3. Endoscopic myotomy is carried out in a proximal to distal direction to a total length more than 7 cm. The expected end point of myotomy is 2 cm distal to the GEJ.
  4. Myotomy of inner circular muscle bundles and outer longitudinal muscle layer is done.
  5. Closure of mucosal entry: the mucosal incision is closed using hemostatic clips.
  Arms: full-thickness myotomy
Procedure: circular myotomy — 1. Entry to submucosal space. After submucosal injection, a 2-cm longitudinal mucosal incision is made at approximately 8-10 cm proximal to the gastroesophageal junction (GEJ).
  2. Submucosal tunnelling. A long submucosal tunnel is created to 3 cm distal to the GEJ.
  3. Endoscopic myotomy is carried out in a proximal to distal direction to a total length more than 7 cm. The expected end point of myotomy is 2 cm distal to the GEJ.
  4. Myotomy of inner circular muscle bundles is done, leaving the outer longitudinal muscle layer intact.
  5. Closure of mucosal entry: the mucosal incision is closed using hemostatic clips.
  Arms: circular myotomy

SUMMARY:
This study compares the clinical efficacy of safety of circular myotomy and full-thickness myotomy guided by peroral endoscopic in treatment of incision length of ≤7cm and of ≥7cm in achalasia patients.

DETAILED DESCRIPTION:
Esophageal achalasia is an esophageal motor disorder, which is characterized by the absence of esophageal peristalsis combined with a defective relaxation of the lower esophageal sphincter (LES). The major symptoms of esophageal achalasia are dysphagia, chest pain, and regurgitation of undigested food.

Currently, treatment options mainly focus on relief of the symptoms by reducing the LES pressure. Pneumatic dilation is the main endoscopic therapies for esophageal achalasia. However, the patients need repeat treatment to maintain therapeutic success and there is a risk of perforation (1%-3%). For surgery approaches, the laparoscopic Heller's myotomy (LHM) combined with Dor's antireflux procedure has gained considerable interest. The LHM can sustain therapeutic effects for long-term in approximately 80% of patients.

Recently, Inoue et al. succeeded in treating achalasia endoscopically with a method called peroral endoscopic myotomy (POEM) and achieved promising results in short-term. Technically, POEM derived from natural orifice transluminal endoscopic surgery (NOTES) and endoscopic submucosal dissection (ESD), in which a submucosal tunnel is created after submucosal injection, and then an endoscopic myotomy was made at the gastroesophageal junction.

However, the clinical efficacy of safety of circular myotomy and full-thickness myotomy guided by peroral endoscopic in treatment of incision length of ≤7cm and of ≥7cm in achalasia patients were not determined, and there was no prospective study that compared different surgical procedures of POEM for esophageal achalasia. Therefore, we aim to compare the clinical efficacy of safety of circular myotomy and full-thickness myotomy guided by peroral endoscopic in treatment of incision length of ≤7cm and of ≥7cm in achalasia patients.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 75 years of age;
2. Patient with esophageal achalasia;
3. Eckardt score > 3;
4. Signed informed consent.

Exclusion Criteria:

1. Severe cardio-pulmonary disease or other serious disease leading to unacceptable surgical risk;
2. Pseudo-achalasia, Mega-oesophagus (greater than 7 cm), or Oesophageal diverticula in the distal oesophagus;
3. Previous endoscopic Botox injection;
4. Previous oesophageal or gastric surgery;
5. Pregnancy or lactation women, or ready to pregnant women;
6. Not capable of filling out questionnaires.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-12; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Therapeutic success | From date of randomization until the follow-up ended, assessed up to 5 years
  Therapeutic success is defined as a symptom control to an Eckardt score of 3 or less. The Eckardt score is the sum of the symptom scores for dysphagia, regurgitation, and chest pain (with a score of 0 indicating the absence of symptoms, 1 indicating occasional symptoms, 2 indicating daily symptoms, and 3 indicating symptoms at each meal) and weight loss (with 0 indicating no weight loss, 1 indicating a loss of <5 kg, 2 indicating a loss of 5 to 10 kg, and 3 indicating a loss of >10 kg) (Eckardt, V. Gastroenterology, 1992. 103(6): p. 1732-8.)

SECONDARY OUTCOMES:
Procedure related complication | From date of randomization until the follow-up ended, assessed up to 5 years
  Perforation, Delayed bleeding, Pneumothorax, Subcutaneous emphysema, Anastomotic leak etc.
Time of treatment failure | From date of randomization until the follow-up ended, assessed up to 5 years
  Time of treatment failure is defined as when the Eckardt score of patients are more than 3.
Pressure at the lower esophageal sphincter | From date of randomization until the follow-up ended, assessed up to 5 years
  From date of randomization until the follow-up ended, assessed up to 5 years
Quality of life | From date of randomization until the follow-up ended, assessed up to 5 years
  Patients will complete the quality-of-life questionnaires (the Medical Outcomes Study 36-Item Short-Form Health Survey, SF-36) for assessing quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Gong, Doctor, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Inoue H, Minami H, Kobayashi Y, Sato Y, Kaga M, Suzuki M, Satodate H, Odaka N, Itoh H, Kudo S. Peroral endoscopic myotomy (POEM) for esophageal achalasia. Endoscopy. 2010 Apr;42(4):265-71. doi: 10.1055/s-0029-1244080. Epub 2010 Mar 30. PMID 20354937
- [Background] Boeckxstaens GE, Annese V, des Varannes SB, Chaussade S, Costantini M, Cuttitta A, Elizalde JI, Fumagalli U, Gaudric M, Rohof WO, Smout AJ, Tack J, Zwinderman AH, Zaninotto G, Busch OR; European Achalasia Trial Investigators. Pneumatic dilation versus laparoscopic Heller's myotomy for idiopathic achalasia. N Engl J Med. 2011 May 12;364(19):1807-16. doi: 10.1056/NEJMoa1010502. PMID 21561346
- See also: Homepage of Nanfang Hospital of Southern Medical University — http://www.nfyy.com/
- See also: Homepage of Department of Gastroenterology, Nanfang Hospital of Southern Medical University — http://www.xhbnet.com/